CLINICAL TRIAL: NCT07146061
Title: Partial Cardiac Denervation to Prevent POAF After CABG: 3 Year Follow-up of pCAD-POAF Randomized Trial
Brief Title: pCAD-POAF 3 Year Follow-up
Status: Not yet recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025-GSP-GG-12
Record Dates: First submitted 2025-08-14; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease; Atrial Fibrillation
Keywords: coronary artery disease; atrial fibrillation
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: This group underwent partial cardiac denervation procedure as well as CABG in the pCAD-POAF trial. However, no other intervention was performed after completing the pCAD-POAF trial.
  Interventions: Other: no other intervention
- Control group: This group only underwent CABG in the pCAD-POAF trial. Likewise, no other intervention was performed after completing the pCAD-POAF trial
  Interventions: Other: no other intervention

INTERVENTIONS:
Other: no other intervention — This is a observational study.

SUMMARY:
This study will include the subjects who enrolled in pCAD-POAF trial (NCT05009914) to observe clinical outcomes 3 years after surgery.

The primary outcome is the AF burden during 3-day continuous ECG monitoring among 2 groups in pCAD-POAF trial 3 years after surgery.

The secondary outcomes are：1. Freedom of AF without the use of antiarrhymic medications or interventions ; 2. The occurence of MACCE (including all-cause mortality, stroke, myocardial infarction, systemic arterial embolism, revascularization, and rehospitalization for heart failure); 3. AF incidence in 3 years and recorded by continuous ECG monitoring; 4. Post-operative antiarrhythmic interventions and occurrence of arrhythmias other than AF; 5. The mean, maximum, and minimum heart rate recorded by Holter monitoring, as well as heart rate variability (HRV); 6. Quality of life assessment, such as EQ-5D-5L and AFEQT.

DETAILED DESCRIPTION:
This study aimed to observe clinical outcomes 3 years after surgery in patients enrolled in pCAD-POAF trial.

After completing the pCAD-POAF trial, investigators would not make any other interventions on enrolled patients. At the 3 year follow-up visit, all subjects will undergo regular laboratory test , electrocardiogram (ECG), ultrasound cardiography (UCG). Besides, coronary computed tomographic angiography(CCTA) will be performed depending on their own willingness. In the meantime, all subjects will be continuously monitored by wearing specific device for the detection of arrhythmias. Data collection will also include the use of medications, medical tests, any documented arrhythmias and the occurrence of clinical events within the 3 years.

In conclusion, this is a extensive follow-up of previous RCT and a non-interventional, observational study.

ELIGIBILITY:
Inclusion Criteria:

* This study will include the subjects who enrolled in pCAD-POAF trial

Exclusion Criteria:

* This study will include the subjects who enrolled in pCAD-POAF trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population enrolled previously in pCAD-POAF trial.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
AF burden | 3 year after the surgery
  the AF burden during 3-day continuous ECG monitoring among 2 groups at the 3 year follow-up.

SECONDARY OUTCOMES:
Freedom of AF without the use of antiarrhymic medications or interventions | within 3 year after surgery
  Freedom of AF without the use of antiarrhymic medications or interventions
The occurence of MACCE | within 3 year after surgery
  including all-cause mortality, stroke, myocardial infarction, systemic arterial embolism, revascularization, and rehospitalization for heart failure
AF incidence in 3 years and recorded by continuous ECG monitoring | 3 year after the surgery
  AF incidence in 3 years and recorded by continuous ECG monitoring
Post-operative antiarrhythmic interventions and occurrence of arrhythmias other than AF | within 3 year after surgery
  Post-operative antiarrhythmic interventions and occurrence of arrhythmias other than AF
The mean, maximum, and minimum heart rate and HRV | 3 year after the surgery
  recorded by Holter monitoring at the 3 year follow-up visit
Assessment of quality of life | 3 year after the surgery
  Assessed by EQ-5D-5L (EuroQol 5-Dimensions 5-Levels questionnaire, higher score means better outcome) and AFEQT (Atrial-Fibrillation-Effect-on-Quality-of-life-Questionnaire, higher score means better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Wei Feng, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, CAMS & PUMC, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided